CLINICAL TRIAL: NCT05077098
Title: A Phase 1 Study of ADXS-504, a Cancer Type Specific Immunotherapy, With Biochemically Recurrent Prostate Cancer
Brief Title: Study of ADXS-504 Immunotherapy for Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Stein (Other)
Responsible Party: Sponsor-Investigator, Mark Stein, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT0847
Record Dates: First submitted 2021-09-19; First posted 2021-10-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Prostate Cancer
Keywords: Cancer Type Specific Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADXS-504 Monotherapy Dose Escalation (Experimental): Subjects with Biochemically Recurrent Prostate Cancer will receive ADXS-504 with dose escalation schema.
  Interventions: Drug: ADXS-504

INTERVENTIONS:
Drug: ADXS-504 — ADXS-504 will be administered as monotherapy at 2 dose levels. Subjects who are assigned to receive Dose Level 1 (DL1) will be administered ADXS-504 at a dose of 1×107 CFU q4 weeks (±3 days) from Week 1 to Week 21. Subjects who are assigned to receive Dose Level 2 (DL2) will be administered ADXS-504 at a dose of 1×108 CFU q4 weeks (±3 days; Week 1 to Week 21). All 3-6 subjects must be enrolled in DL1, and DL1 must be confirmed safe, before enrollment for DL2 may begin. For both dose levels, these doses are followed by maintenance dosing at each respective dose level given every 12 (q12) weeks (±3 days) for 4 doses for overall total of 10 doses of the study treatment. If DL1 is deemed to exceed the MTD, dose reduction of ADXS-504 to DL-1 (1×106 CFU) may proceed. Dose level -1, intermediate dose levels or expansion of a cohort may also be further evaluated if recommended by the Investigator and Advaxis in future amendments.
  Other Names: ADXS-504 immunotherapy

SUMMARY:
Primary Objective:

- To evaluate the safety and tolerability of ADXS-504 and to determine the MTD (maximum tolerated dose) or RP2D (recommended phase two dose)

Secondary Objectives:

* To characterize the immunological activity of ADXS-504, administered as; and to characterize the genomic profiles of study subjects
* To evaluate the effects of ADXS-504 on change in PSA
* To evaluate time to PSA progression

DETAILED DESCRIPTION:
ADXS-504 is a novel Listeria monocytogenes (Lm) - based immunotherapy, bioengineered to elicit T cell responses against 24 tumor antigens that include 1) 14 peptide antigens derived from frequently occurring and commonly shared hotspot mutations in patients with prostate cancer and 2) 10 peptide antigens derived from sequence-optimized tumor associated antigens (TAAs) that are differentially expressed or overexpressed in prostate cancer. ADXS-504 is designed to express multiple tumor antigen targets to which patients may generate a broad set of effector T cells for tumor control.

This is a phase 1 open-label study of ADXS-504 monotherapy in subjects with biochemically recurrent prostate cancer previously treated with radical prostatectomy (RP) or radiation therapy (external beam or brachytherapy) who are not currently receiving androgen ablation therapy. The purpose of this study is to evaluate safety, tolerability, and preliminary clinical and immune responses following treatment with ADXS-504 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Histologically documented prostatic adenocarcinoma confirmed by a pathology report from prostate biopsy or a radical prostatectomy specimen.
2. Age ≥18 years
3. Previously undergone primary therapy for prostate cancer. Salvage XRT or cryotherapy following primary therapy ≥ 6 months prior to randomization is allowed.
4. A rising prostate specific antigen (PSA) defined as the following

   * If the subject's primary therapy was radical prostatectomy (RP) (with or without adjuvant or salvage XRT), rising PSA is defined as 2 consecutive rising values above 0.1 ng/mL, each taken ≥ 3 weeks apart, and the last value ≥ 0.3 ng/mL
   * If the subject received other primary therapies (e.g. XRT, cryosurgery, brachytherapy), rising prostate specific antigen (PSA) is defined per the Phoenix definition, i.e., 2 consecutive rising values above the PSA nadir plus 2.0 ng/mL.
5. PSA ≥0.3 in addition to prostate-specific antigen doubling time (PSADT)≥4 months. PSADT will be determined from all non-zero PSA values within 12 months prior to registration. To calculate PSADT, there must be at least THREE PSA values, with at least 3 weeks between each measurement. The PSADT will be computed from the formula: PSADT = (loge2)/k, with k being the estimated slope of the logarithm of PSA over time.

   The following web site may also be used:

   http://www.mskcc.org/applications/nomograms/prostate/PsaDoublingTime.aspx
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, or Karnofsky score ≥ 70%
7. Testosterone ≥ 150 ng/dL ≤ 28 days of prior to registration
8. Adequate bone marrow, hepatic, and renal function.
9. Subject has baseline blood oxygen saturation on room air of ≥95%;
10. Subject has the ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures
11. Subject is willing and able to provide an archived biopsy specimen which may be used for correlative studies and to determine human leukocyte antigen(HLA) type;
12. Subject with a female partner of child-bearing potential is eligible if he agrees to follow the contraceptive guidance, provided in Appendix 5, during the treatment period and for at least 120 days after the final dose of study treatment.

Exclusion Criteria:

Medical Conditions

1. Subject has evidence of measurable or evaluable metastatic disease on bone or computed tomography (CT) or positron emission tomography(PET) scans performed ≤8 weeks of registration (patients with PET scan findings consistent with metastasis but who have normal conventional imaging by CT/MRI/Bone scan using standard radiographic criteria ARE eligible)
2. Subject has known brain metastasis. Subjects with neurological symptoms must undergo a CT scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis;
3. Subject has an active autoimmune disease requiring systemic treatment within the past 3 months, a documented history of clinically severe autoimmune disease, or a disorder that requires systemic corticosteroids or immunosuppressive agents. Subjects with vitiligo, psoriasis, alopecia or resolved childhood asthma/atopy not requiring systemic treatment would be an exception to this rule. Subjects with hypothyroidism who are stable on hormone replacement (>10 mg daily prednisone equivalent) or Sjögren's syndrome will not be excluded from the study;
4. Subject has had an allogeneic tissue/solid organ transplant;
5. Subject has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies);
6. Subject has a known active hepatitis B (e.g., hepatitis B virus surface antigen reactive) or hepatitis C infection (e.g., hepatitis C virus RNA [qualitative] is detected);
7. Subject has an active infection requiring systemic therapy or is dependent on or currently receiving antibiotics that cannot be discontinued before dosing. (Note: Subjects who discontinue an antibiotic prior to dosing must wait at least 5 half-lives after the last dose of antibiotic before receiving any study treatment);
8. Subject has an implanted medical device that poses a high risk for bacterial colonization and/or that cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screws, metal plates, bone grafts, or other exogenous implants). NOTE: More common devices and prosthetics that include arterial and venous stents, dental and breast implants and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device or implant;
9. Subject has a contraindication (e.g., sensitivity/allergy) to trimethoprim/ sulfamethoxazole; ampicillin; ciprofloxacin
10. Subject has a contraindication to NSAIDs;
11. Subject has a known allergy to any component of the study formulation(s);
12. Subject has a history of listeriosis;
13. Subject has had a major surgery, open biopsy or significant traumatic injury ≤6 weeks of registration;
14. Subject has any other serious or uncontrolled physical or mental condition/disease that, as judged by the Investigator, could place the subject at higher risk derived from their participation in the study, could confound results of the study, or would be likely to prevent compliance with the requirements of the study.
15. Subject has a second primary malignancy with greater than minimal metastatic potential that has not been in remission for greater than 3 years. Examples of tumors that do not require a 3-year remission: non-melanoma skin cancer, resected melanoma in situ, or non-muscle invasive urothelial carcinoma.

Prior/Concomitant Therapy

1. Subject is on or has received Luteinizing hormone-releasing hormone (LHRH) agonists, LHRH antagonists within 6 months prior to study enrollment;
2. Subject has received oral antiandrogens within 3 months prior to study enrollment;
3. Subject has received agents such as 5 alpha reductase inhibitors, ketoconazole, megestrol acetate, systemic steroids, or herbal supplements that are known to affect PSA (PC-SPES, saw palmetto oil) within the past month;

   Prior/Concurrent Clinical Study Experience
4. Subject is currently participating in or has participated in a study of an investigational agent(s) within 4 weeks of the first dose of study treatment;

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of adverse events (AEs), graded by CTCAE v 5.0 (Common Terminology Criteria for Adverse Events) | 28 days
  To determine safety and tolerability profile of ADXS-504 of the investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No